CLINICAL TRIAL: NCT06968039
Title: This Study is Designed to Evaluate the Efficacy of Personalized Alternating Current Stimulation in the Treatment of Working Memory in Patients With Inflammatory Demyelination of the Central Nervous System
Brief Title: Effectiveness of Personalized Alternating Current Stimulation for Treating Cognitive Impairment in CNS Demyelination Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xw-tES-04
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Electric Stimulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromodulation Group (Experimental)
  Interventions: Device: Neuroelectrics StarStim 32
- Sham Neuromodulation Group (Sham Comparator)
  Interventions: Device: Neuroelectrics StarStim 32

INTERVENTIONS:
Device: Neuroelectrics StarStim 32 — Using the advanced Neuroelectrics StarStim 32 device from Spain, individualized imaging modeling systems are employed to precisely target the frontal and parietal cortex. Personalized EEG-guided electrical stimulation protocols are selected. The stimulation parameters are as follows: a current intensity of 2 mA, a duration of 21 minutes per session for one time with EEG monitoring conducted before and after electrical stimulation.
  Arms: Neuromodulation Group
Device: Neuroelectrics StarStim 32 — Sham stimulation is performed using the same device and procedures as the neuromodulation group. The stimulator automatically shuts off after 30 seconds, while maintaining the device's connection. This design creates an initial sensation similar to actual stimulation while preserving the double-blind nature of the study.
  Arms: Sham Neuromodulation Group

SUMMARY:
Background: Central nervous system inflammatory demyelinating diseases often lead to significant cognitive impairment, presenting a critical challenge in patient management.

Objective: To evaluate the effectiveness of individualized transcranial electrical stimulation (tES) in improving cognitive function among patients with inflammatory demyelinating disorders.

Methods: This study will assess cognitive performance through standardized neuropsychological assessments before and after individualized a one-time tES intervention, measuring changes in cognitive domains including working memory, attention, executive function, and processing speed.

Anticipated Results: We hypothesize that personalized transcranial electrical stimulation will demonstrate significant improvements in cognitive performance, potentially offering a non-invasive therapeutic approach for managing cognitive decline in central nervous system inflammatory demyelinating diseases.

Significance: This research may provide novel insights into neuromodulation strategies for cognitive rehabilitation in patients with complex neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Neuromyelitis Optica Spectrum Disorders (NMOSD), Multiple Sclerosis (MS), and other Central Nervous System Inflammatory Demyelinating Diseases that meet diagnostic criteria;
* Patients with SDMT scores <55 or subjective cognitive decline;
* Age between 18 and 65 years, gender unrestricted;
* No relapse or medication changes in the past month;
* EDSS (Expanded Disability Status Scale) score ≤6;
* Right-handed, native Chinese speakers with sufficient educational background to understand the test instructions; -Willing to participate and have signed informed consent.-

Exclusion Criteria:

* Relapse record within the past month;
* Medication adjustment within the past month or having undergone modified electroconvulsive therapy, transcranial magnetic stimulation, or other neuromodulation techniques;
* Participating in any other clinical research within 1 month prior to enrollment or currently;
* Presence of cochlear hearing aids, cardiac pacemakers, or implanted brain stimulation devices;
* Skin integrity damage at electrode placement sites, or allergy to electrode gel or adhesives;
* History of epilepsy, hydrocephalus, central nervous system tumors, brain injury, or intracranial infections;
* Pregnant or lactating women, or those planning pregnancy in the near future;
* Scoring ≥3 on item 3 (suicide item) of the HDRS-17 or concurrent severe mental illness;
* Concurrent severe or unstable organic diseases;
* Unable to cooperate with treatment, follow-up, or clinical, EEG, and imaging data collection due to poor patient compliance;
* Other situations deemed inappropriate for study participation by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Working Memory Training-Related Scores | An hour before and after interventions
  Working Memory Related Task is a widely used paradigm in cognitive psychology and neuroscience to study memory retention and recognition. In this task, participants are first presented with a image stimulus for a brief period. After a delay interval, they are shown a set of test stimuli, including the original sample and one or more distractors. The participants' task is to identify whether the sample stimulus is present among the test items. This paradigm allows researchers to investigate the effects of delay duration on memory accuracy and the neural mechanisms underlying memory encoding, maintenance, and retrieval.
SDMT (Symbol Digit Modalities Test) | An hour before and after interventions.
  The SDMT is a widely used test to measure processing speed and cognitive flexibility. Participants are asked to match symbols with corresponding numbers according to a key, which they must do as quickly as possible. This task assesses visual scanning, motor speed, and the ability to shift attention.

SECONDARY OUTCOMES:
AVLT (Auditory Verbal Learning Test) | Before interventions
  The AVLT is a neuropsychological test used to assess verbal memory. It involves presenting a list of words to participants, who are then required to recall the words immediately after presentation and after a delay. The test examines both short-term and long-term verbal memory retention, as well as the ability to organize and retrieve information.
Digit Span Test | An hour before interventions
  The Digit Span test measures working memory and attention. Participants are presented with a sequence of digits, and they must repeat the sequence either in the same order (forward span) or in reverse order (backward span). The test assesses both short-term memory and cognitive flexibility.
BVMTR (Brief Visual Memory Test-Revised) | An hour before and after interventions.
  The BVMTR is designed to evaluate visual memory and recognition. Participants are shown a set of geometric shapes, which they must remember. After a delay, they are asked to identify which shapes were previously shown among distractors. This test helps in assessing visual memory and the ability to recognize visual stimuli.
STROOP (Stroop Color and Word Test) | An hour before and after interventions.
  The Stroop test assesses cognitive flexibility and the ability to inhibit automatic responses. Participants are presented with words printed in different ink colors and must name the ink color rather than reading the word itself (which can be incongruent). The task evaluates cognitive control, selective attention, and response inhibition.

OTHER OUTCOMES:
EDSS (Expanded Disability Status Scale) | At baseline.
  The EDSS is a scale used to measure the severity of disability in multiple sclerosis (MS) patients. It assesses both neurological impairment and physical function through a series of clinical examinations, including motor function, sensory function, coordination, and cognitive ability.
MFIS (Modified Fatigue Impact Scale) | At baseline
  The MFIS is a self-report questionnaire used to assess the impact of fatigue on daily functioning. It consists of questions about physical, cognitive, and psychosocial functioning, measuring how fatigue affects different areas of a person's life.
MSIS (Multiple Sclerosis Impact Scale) | At baseline
  The MSIS is a questionnaire designed to measure the impact of multiple sclerosis on a patient's physical and psychological well-being. It includes questions about physical disability, mobility, fatigue, and emotional well-being, providing an overall assessment of the disease's impact on quality of life.
HAMA (Hamilton Anxiety Rating Scale) | At baseline
  The HAMA is a clinician-administered scale used to assess the severity of a patient's anxiety. It includes 14 items that evaluate both psychological and physical symptoms of anxiety, such as tension, fear, and physiological symptoms (e.g., palpitations).
HAMD (Hamilton Depression Rating Scale) | At baseline
  The HAMD is a clinician-administered scale that assesses the severity of depression symptoms. It includes 17 items that evaluate mood, behavior, and physical symptoms, such as sleep disturbances, appetite changes, and guilt.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No